CLINICAL TRIAL: NCT05919511
Title: A Prospective, Observational Cohort Study of Participants at Risk for Chronic Graft-Versus-Host Disease in the United States (THRIVE)
Brief Title: Observational Study for Patients at Risk for Chronic Graft-Versus-Host Disease
Acronym: THRIVE
Status: Recruiting | Type: Observational
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-GVHD-401
Record Dates: First submitted 2023-05-05; First posted 2023-06-26 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: cGVHD
Keywords: chronic graft versus host disease; cGVHD; MA-GVHD-401; THRIVE; GVHD; chronic GVHD; allogenic stem cell transplant (alloSCT)
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- At risk for GVHD: Equal or Greater than 18 years old post alloSCT
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — This is an observational study

SUMMARY:
The purpose of this prospective observational study is to collect data from participants who have recently had an allogenic Stem Cell Transplant(alloSCT) and are at risk of Chronic Graft Versus Host Disease(cGVHD)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years inclusive at the time of signing the ICF
* Allogeneic SCT 90 to 180 days prior to enrollment
* Able to comprehend and willing to provide informed consent
* Willing and able to complete participant-assessment questionnaires either alone or with minimal assistance from a caregiver and/or trained site personnel

Exclusion Criteria:

* There are no exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants greater than or equal to 18 years of age who have had Allogenic SCT 90 to 180 days prior to enrollment
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Overall Burden of cGVHD diagnosis and severity | 36 months

SECONDARY OUTCOMES:
To describe personal and healthcare resources associated with the management of cGVHD | 36 months
To describe changes in the proteomic, cytologic and molecular profile in blood, serum and saliva cGVHD | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - City of Hope, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Moffit Cancer Center, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Cancer Center, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Group, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - Tulane Cancer Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts Cancer Research Center, Boston, Massachusetts
  - Corewell Health, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Geisinger Health Systems, Danville, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Observational Study for Patients at Risk for Chronic Graft-Versus-Host Disease (THRIVE) — https://www.incyteclinicaltrials.com/study/?id=MA-GVHD-401&SearchTerm=MA-GVHD-401&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=